CLINICAL TRIAL: NCT03932877
Title: An Analysis Soluble Endoglin and Matrix Metalloproteinase 14 With Elisa Method in the Diagnosis and Severity of Early/Late-onset Preeclampsia
Brief Title: Serum Soluble Endoglin and Matrix Metalloproteinase 14 With Elisa Method in Early/Late-onset Preeclampsia
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH3
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Matrix Metalloproteinase 14

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- late-onset preeclampsia, group1: 30 late-onset preeclampsia patients as group1 (gestational age≥34 weeks). The diagnosis of preeclampsia, as defined by the Committee on Terminology of the American College of Obstetricians and Gynecologists (ACOG), will establish based on the presence of proteinuria (urinary excretion of 300 mg protein or higher, or at least 1+in dipstick in a 24-h urine specimen) and a blood pressure level of ≥140/90mmHg (two blood pressure measurements 6 h apart) that occurs after 20 weeks of gestation in a previously normotensive woman. Diastolic and/or systolic blood pressure up to 110/160 mm Hg will consider mild, and higher values will consider to being severe.
  Interventions: Other: MMP-14 and s-ENG levels
- Control, group 2: 33 patients with normal pregnancies as group2 (gestational age≥34 weeks). The control groups' samples obtained during the routine obstetrical care examination in the third trimester of pregnancy. Then these pregnant women followed-up until the delivery.
  Interventions: Other: MMP-14 and s-ENG levels
- early-onset preeclampsia, group 3: 31 early-onset preeclampsia patients as group3 (gestational age<34 weeks). The diagnosis of preeclampsia, as defined by the Committee on Terminology of the American College of Obstetricians and Gynecologists (ACOG), will establish based on the presence of proteinuria (urinary excretion of 300 mg protein or higher, or at least 1+in dipstick in a 24-h urine specimen) and a blood pressure level of ≥140/90mmHg (two blood pressure measurements 6 h apart) that occurs after 20 weeks of gestation in a previously normotensive woman. Diastolic and/or systolic blood pressure up to 110/160 mm Hg considered mild, and higher values considered to being severe.
  Interventions: Other: MMP-14 and s-ENG levels
- Control, group 4: 31 patients with normal pregnancies as group 4 (gestational age<34 weeks). The control groups' samples obtained during the routine obstetrical care examination in the third trimester of pregnancy. Then these pregnant women followed-up until the delivery.
  Interventions: Other: MMP-14 and s-ENG levels

INTERVENTIONS:
Other: MMP-14 and s-ENG levels — Venous blood sampled from the antecubital veins for measuring the serum concentration of MMP-14 and s-ENG levels. The serum MMP-14 and s-ENG levels measured using commercially available reagent kits, which is produced to detect human MMP-14 and s-ENG levels (Rel Assay Diagnostics Gaziantep, Turkey). The MMP-14 and s-ENG levels measurements were performed in accordance with the company's protocol.

SUMMARY:
Objective: Defective placentation and inadequate trophoblastic invasion have an important place in the aetiology of preeclampsia (PrE). Trophoblasts invade the maternal decidua and remodel spiral arteries with matrix metalloproteinase-14 (MMP-14). To the best of our knowledge, studies of MMP-14 protein levels of PrE patients' sera remain unpublished. This study aims to investigate the value of serum MMP-14 and soluble endoglin (s-ENG) in PrE patients and healthy controls.

Methods: The study was conducted with 30 late-onset preeclampsia patients (L-PrE) as group1 (gestational age≥34 weeks), 33 patients with normal pregnancies as group2 (gestational age≥34 weeks), 31 early-onset preeclampsia patients (E-PrE) as group3 (gestational age<34 weeks), and 31 patients with normal pregnancies as group 4 (gestational age<34 weeks). Serum MMP-14 and s-ENG levels measured by ELISA were compared.

DETAILED DESCRIPTION:
The study was conducted at Cengiz Gokcek Women's and Children's Hospital, Gaziantep, Turkey at department of obstetrics and gynecology between date of January 2018 and December 2018. The study protocol was designed according to the Declaration of Helsinki, and the institutional ethical review board of Gaziantep University approved the study (Reference number: 2018/91). One hundred twenty-five women enrolled in the study in four groups. The investigators consecutively recruited 61 pregnancies complicated with preeclampsia, and 64 healthy pregnancies will select for the control group. All participiants gave their oral and written informed consent before their inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia
* healthy pregnancy

Exclusion Criteria:

* pregnant women with any systemic condition (such as chronic hypertension, diabetes mellitus, thyroid diseases, liver and kidney diseases)
* women with a history of drug use throughout pregnancy
* history of medication for PE treatment at the time of first admission
* patients who had fetal congenital abnormalities or genetic syndromes
* multiple gestations
* active labour

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy. Preeclampsia is a pregnancy complication characterized by high blood pressure and signs of damage to another organ system, most often the liver and kidneys. Preeclampsia usually begins after 20 weeks of pregnancy in women whose blood pressure had been normal. Early-onset preeclampsia is usually defined as preeclampsia that develops before 34 weeks of gestation, whereas late-onset preeclampsia develops at or after 34 weeks of gestation.
Study Population: The investigators consecutively will recruite 61 subjects with preeclampsia, and 64 healthy preganancies will selecte for the control group.
  Preeclampsia is a pregnancy complication characterized by high blood pressure and signs of damage to another organ system, most often the liver and kidneys. Preeclampsia usually begins after 20 weeks of pregnancy in women whose blood pressure had been normal. Early-onset preeclampsia is usually defined as preeclampsia that develops before 34 weeks of gestation, whereas late-onset preeclampsia develops at or after 34 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Serum matrix metalloproteinase-14 levels in preeclampsia | 1 day
  The primary endpoint in this analysis is to evaluate the value of serum matrix metalloproteinase-14 levels (ng/ml) in preeclampsia patients and also address its relationship with its severity.

SECONDARY OUTCOMES:
Serum soluble endoglin levels in preeclampsia | 1 day
  The secondary endpoint in this analysis is to evaluate the value of serum soluble endoglin levels (ng/ml) in preeclampsia patients and also address its relationship with its severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ovayolu, Principal Investigator — Cengiz Gokcek WCH
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhang XH, Zhang HY, Lu S, Jiang LL, Wu J, Yang YL, Zhang SA. MMP-14 aggravates onset of severe preeclampsia by mediating soluble endoglin release. Eur Rev Med Pharmacol Sci. 2018 Mar;22(5):1209-1215. doi: 10.26355/eurrev_201803_14460. PMID 29565476
- [Result] Espino Y Sosa S, Flores-Pliego A, Espejel-Nunez A, Medina-Bastidas D, Vadillo-Ortega F, Zaga-Clavellina V, Estrada-Gutierrez G. New Insights into the Role of Matrix Metalloproteinases in Preeclampsia. Int J Mol Sci. 2017 Jul 20;18(7):1448. doi: 10.3390/ijms18071448. PMID 28726716
- [Result] Kaitu'u-Lino TJ, Palmer KR, Whitehead CL, Williams E, Lappas M, Tong S. MMP-14 is expressed in preeclamptic placentas and mediates release of soluble endoglin. Am J Pathol. 2012 Mar;180(3):888-894. doi: 10.1016/j.ajpath.2011.11.014. Epub 2012 Jan 31. PMID 22296769
- [Derived] Ovayolu A, Karaman E, Turgut A, Cekici Y, Ortabag T, Chiara Rapisarda AM, Noventa M, Cianci A. Endothelial cell-specific-molecule-1 (endocan) levels in women with premature ovarian insufficiency: a prospective comparative study. J Obstet Gynaecol. 2021 May;41(4):637-641. doi: 10.1080/01443615.2020.1789952. Epub 2020 Aug 18. PMID 32808833

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03932877/Prot_SAP_000.pdf